CLINICAL TRIAL: NCT01221116
Title: Inotropic Treatment With Levosimendan (SimdaxR)in Heart Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to difficulties in including patients
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Ullevaal University Hospital, Knut Arvid Kirkebøen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INSI-study
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2003-01

CONDITIONS: Heart Failure; Cardiac Surgery
Keywords: coronary artery disease,; aortic stenosis,; heart failure
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease; Aortic Valve Stenosis | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1: Type of surgery (No Intervention): Two types of patients are compared (placebo vs levosimendan): CABG - coronary artery bypass grafting and AVR - aortic valve replacement (either with or without CABG - coronary artery bypass grafting)
  Interventions: Drug: levosimendan

INTERVENTIONS:
Drug: levosimendan — levosimendan 0.1 microgram/kg/min) for 24 hours
  Other Names: Type of surgery

SUMMARY:
Hypothesis: Treatment with levosimendan will preserve myocardial function and hemodynamics after cardiac surgery and lead to reduced stay at intensive care unit

DETAILED DESCRIPTION:
Single center, prospective, randomized parallel-group, double-blinded study

ELIGIBILITY:
Inclusion Criteria:

* EF (ejection fraction)<40%

Exclusion Criteria:

* renal failure, liver failure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Need for inotropic agents or IABP (intra aortal balloon pump) | jan 2003 - dec 2008

SECONDARY OUTCOMES:
Biochemical, echocardiographic data, Gated SPECT (single photon emission gated tomography) data, laser Doppler data, 24 hour ECG (electrocardiogram) data and clinical "all round" data. | jan 2003-dec 2008

CONTACTS AND LOCATIONS:
Overall Officials: Knut A Kirkebøen, MD, PhD, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Dept. of Cardiothoracic Anesthesia, Ullevål University Hospital, Oslo, Oslo County, Norway